CLINICAL TRIAL: NCT05527080
Title: Development of Motility and Cognition in Infants
Acronym: PILKE
Status: Recruiting | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); Aalto University (Other); Tampere University (Other)
Responsible Party: Principal Investigator, Sampsa Vanhatalo, professor in clinical neurophysiology, Helsinki University Central Hospital
Other Study IDs: PILKE
Record Dates: First submitted 2022-08-23; First posted 2022-09-02 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Neurodevelopmental Disorders; Developmental Delay; Development, Infant; Child Development; Cognitive Developmental Delay; Neurophysiologic Abnormality
Keywords: wearable; medical wearable; human activity recognition; growth chart; neurodevelopment
MeSH Terms: conditions — Neurodevelopmental Disorders; Learning Disabilities | interventions — Physical Therapy Modalities; Braces; Casts, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- typically developing infants: recruitment at 5-8mos of age; infants are considered typically developing if they are born at term age with no neurologically significant medical history, and they are not medically followed up for a suspicion of such. The benchmark for this is taken from the nationally harmonized pre/postnatal screening practise.
- neurodevelopmental concern: recruitment at 5-8mos of age; infants are recruited from the outpatient clinic in the New Children's hospital (NCH). They have either a known perinatal risk factor (e.g.stroke, HIE, meningitis), or they are referred to pediatric neurologists at NCH due to a suspected delay or deviance in neurodevelopment.
  Interventions: Other: physiotherapy
- hip dysplasia concern: recruitment at 2-6 weeks of age after perinatal clinical suspicion of hip dysplacia. These infants may be left out of follow-up (mild), or treated by orthopedic clinic with a soft brace (moderate) or a stronger cast (sever)
  Interventions: Device: brace

INTERVENTIONS:
Other: physiotherapy — Some infants will receive physiotherapy as a part of their clinically indicated care.
  Groups: neurodevelopmental concern
Device: brace — Some infants in the hip dysplasia group will receive brace and/or cast as a part of their clinically indicated care
  Other Names: cast
  Groups: hip dysplasia concern

SUMMARY:
PILKE study uses wearables for assessing motor development in infants in order to define functional growth trajectories in the normal infants and infants at risk of neurological compromise. In addition, PILKE studies correlation of early motor development to later neurocognitive development.

DETAILED DESCRIPTION:
PILKE study builds on the recent development of an infant wearable, MAIJU, a multisensor garment that can be used to quantify infants posture and movement patterns out-of-hospital. The study will recruit typically developing infants (control group) and infants with an identified or suspected risk of neurodevelopmental compromise, as well as infants undergoing orthopedic follow-up for hip issues.

Infants will be examined and treated according to clinical routine practise, while MAIJU and other novel measures are added to monitor aspects of neurodevelopment. Recordings with MAIJU will be done every 6-8 weeks from about 5 months to 18 months of age, and the neuropsychological outcome is assessed using Bayley scales at two years of age.

The study is observational by design, and the trajectories of motor performance are compared to other clinically identified measures of development.

ELIGIBILITY:
Inclusion Criteria:

* age at enrollment 5-8mos
* typically developing

Exclusion Criteria:

* all neurologically significant medical histories during pregnancy, at birth or postnatally
* suspicion of developmental delay
* suspicion or diagnosis of syndromes with neuromotor symptoms

Ages: 5 Months to 26 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants at 5-8mos of age. Upper age limit may be extended until the infant learns to stand up.
  Groups have either no medical history (#1) or a suspicion or risk of neurodevelopmental delay/deviance (#2)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
neurocognitive development | 24 months
  The total score of the neuropsychological examination Bayley scales III will be used
neurological development | 12 months
  Binary information (normal vs abnormal) is taken from the postnatal follow-up clinic inspection that is done according to the national standards (www.thl.fi)

CONTACTS AND LOCATIONS:
Overall Officials: Sampsa K Vanhatalo, prof, Principal Investigator — University of Helsinki
Locations (1):
- BABA, Clinical Trial Unit, New Children's Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamada T, Nakamura K, Horie K, Yamashita Y, Iwaku M. [Extent of odontoblast process in normal and carious dentin]. Kokubyo Gakkai Zasshi. 1982 Jun;49(2):325-32. No abstract available. Japanese. PMID 6957504
- [Background] Airaksinen M, Gallen A, Kivi A, Vijayakrishnan P, Hayrinen T, Ilen E, Rasanen O, Haataja LM, Vanhatalo S. Intelligent wearable allows out-of-the-lab tracking of developing motor abilities in infants. Commun Med (Lond). 2022 Jun 15;2:69. doi: 10.1038/s43856-022-00131-6. eCollection 2022. PMID 35721830
- See also: Official study website at the host lab pages — https://www.babacenter.fi/hankkeet/pilke/